CLINICAL TRIAL: NCT02834429
Title: Pre-endoscopy Serological Testing for Coeliac Disease - a Novel Approach Using Rapid Antibody Testing.
Brief Title: Pre-endoscopy Serological Testing for Coeliac Disease; a Novel Approach Using Rapid Antibody Testing
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH15416
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- endoscopy patients: We will recruit patients (n=1000) from the endoscopy department at the Royal Hallamshire Hospital, Sheffield, United Kingdom (UK).

SUMMARY:
The aim of this study is to assess the clinical utility of the whole blood transglutaminase-based rapid test against current serological tests and the gold standard of duodenal biopsy. The investigators will recruit patients (n=1000) from the endoscopy department at the Royal Hallamshire Hospital, Sheffield, United Kingdom (UK). The patients recruited for this study will already have been referred for a consultation and gastroscopy. In addition, these patients will already have been serologically tested for IgA TTG, EMA and a total IgA immunoglobulin level (as per normal clinical practice).

All duodenal biopsy specimens will be fixed in buffered formalin and embedded in paraffin wax. Standard, 3μm thick sections at three levels will be stained with haematoxylin and eosin and reported routinely. Additionally, biopsies demonstrating increased intraepithelial lymphocytes only (changes compatible with but not diagnostic of coeliac disease) will be stained with KiRAS or CD4/CD8 which are markers for coeliac disease.

DETAILED DESCRIPTION:
Coeliac disease is the most common chronic inflammatory bowel condition encountered by physicians. Internationally the prevalence estimated by serological screening in healthy volunteers is between 0.5-1.0%. Historically, patients with adult coeliac disease complained of symptoms suggestive of mal-absorption, diarrhoea, weight loss or anaemia. This manner of presentation is now described as the classical (typical) form. Failure to recognise this disease may be due to the insidious nature of its presentation. Individuals with undiagnosed coeliac disease may have numerous hospital attendances, prior to diagnosis.

Although the presentation of patients with coeliac disease may be protean, serological markers have provided a cheap and non-invasive method by which clinicians in both primary and secondary care can initially recognise patients who may have coeliac disease. The aim of this study is to assess the clinical utility of the whole blood transglutaminase-based rapid test against current serological tests and the gold standard of duodenal biopsy.

Methods:

Study design and Participants Group 1 was a multicentre retrospective analysis of all patients with anaemia attending a gastroscopy with duodenal biopsy at four UK hospitals (Addenbrooke's, Bradford, Hull and Whipps Cross) over a 12 month period ranging from 2012 to 2014. The availability of coeliac serology prior to gastroscopy was reviewed.

Group 2 was a prospective study comparing the sensitivities of Simtomax to conventional serology in an iron deficient cohort. We prospectively recruited 133 consecutive patients (age range: 18-89 years, median 53) with iron deficiency with or without anaemia attending a single coeliac disease research endoscopy list at the tertiary referral centre Royal Hallamshire Hospital between 2013 and 2015. All recruited patients were consented for the study prior to the gastroscopy. The patients concurrently undertook the point-of-care test, Simtomax, conventional coeliac serology (IgA-TTG, IgA-EMA) and total IgA levels at the endoscopy unit. All patients then had a gastroscopy with quadrantic duodenal biopsy from the second part of the duodenum and at least one duodenal bulb biopsy. Patients were excluded from the study if they were known to have coeliac disease or were on a gluten free diet. Patients with coagulopathy, active gastrointestinal bleeding or a suspected carcinoma observed during the examination were also excluded. Clinical information of the patients was available to the endoscopist, however the endoscopist was blinded to the results of the Simtomax test.

Group 3 was a retrospective histological analysis of patients attending a separate non-coeliac specific iron deficiency anaemia clinic at the Northern General Hospital in 2013-2014. We reviewed their duodenal histology and hospital case notes to determine the yield of alternative causes other than coeliac disease in the context of iron deficiency anaemia.

Point-of-care test, Simtomax:

Simtomax is a point-of-care test for coeliac disease manufactured by Augurix Diagnostics, Switzerland. It detects both IgA and IgG antibodies to DGP, as well as the total IgA level. The assay is based on lateral flow immunochromatography using colloidal gold antihuman antibodies as a signal detector. A sample of 25 μl of capillary venous blood is required which can be obtained through a simple finger prick technique. The assay can also be performed using a plasma sample either in ethylenediaminetetraacetic acid (EDTA) or heparin as well as a separated serum sample, although a smaller sample volume of 20 μl is required. The blood sample is then applied to the test device, followed by the application of 5 drops of the provided buffer solution. The result can be read after 10 minutes. Positive results are indicated by the presence of a solid red test line for IgA and/or IgG-DGP positivity. A second single red line indicates the presence of IgA. An in-built red control line ensures a correctly functioning test.

Serology:

Total IgA was measured on a Behring BN2 nephelometer. IgA-TTG antibodies were evaluated using enzyme-linked immunosorbent assay kits (Aesku Diagnostics, Wendelsheim, Germany). An IgA-TTG titre of > 15 U/ml before 20/5/2014, a new cut off level of >9 U/ml from 20/5-11/12/2014, and then >7 U/ml from 12/12/2014 onwards, were regarded as positive as per the manufacturer's guidance. IgA-EMA was detected by immunofluorescence on primate oesophagus sections (Binding Site, Birmingham, UK).

Biopsies and histology

In total, at least five biopsies were taken from the duodenum, including at least one from the duodenal bulb, with each biopsy fixed in formalin at the time of the gastroscopy. Specimens were then processed, orientated and embedded in paraffin wax by the pathology department. Standard 3 µm thick sections at three levels were stained with haematoxylin and eosin, and reported routinely by gastrointestinal histopathologists without knowledge of the Simtomax results. Villous atrophy was graded according to the modified Marsh criteria.

Diagnosis of coeliac disease:

The presence of villous atrophy (Marsh 3a-3c) on histology with a positive IgA-EMA or IgA-TTG were required for the diagnosis of coeliac disease. In cases of seronegative villous atrophy, human leucocyte antigen (HLA) genotyping was performed, with a negative HLA DQ2 or DQ8 phenotype used to rule out coeliac disease. Supporting information such as family history and response to a gluten free diet were also taken into account.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or more undergoing clinically indicated gastroscopy with biopsy and coeliac serology testing

Exclusion Criteria:

* Patients with coagulopathy (INR > 1.3 Platelets < 80)
* Active gastrointestinal bleeding identified at endoscopy
* suspected carcinoma identified at gastroscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Endoscopy patients at the Royal Hallamshire Hospital Sheffield
Sampling Method: Non-Probability Sample
Enrollment: 1596 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Positive and negative predictive values of the whole blood transglutaminase-based rapid test tissue for diagnosing coeliac disease | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: David Sanders, Study Director — Sheffield Teaching Hospitals NHS FT
Locations (1):
- Department of Gastroenterology, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No